CLINICAL TRIAL: NCT06277518
Title: Establishment and Application of Decision System for Postoperative Admission to ICU for Patients With Digestive System Malignancy
Brief Title: System for Postoperative Admission to ICU for Patients With Digestive System Malignancy
Status: Active, not recruiting | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Liqin Deng
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Malignant tumors of digestive system; Intensive care Unit; risk factors; predictive models
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group,: the risk factors of patients with malignant tumors of digestive system meeting the inclusion criteria were observed without special intervention
  Interventions: Procedure: Surgery for malignant tumors of the digestive system

INTERVENTIONS:
Procedure: Surgery for malignant tumors of the digestive system — Related treatment or palliative surgery under general anesthesia for digestive system malignancies

SUMMARY:
Postoperative admission to ICU for patients with digestive system tumors is one of the most common postoperative complications of all non-cardiac surgeries. The study found that supportive treatment of critically ill patients admitted to ICU after surgery was conducive to reducing mortality, and the most common complications of postoperative ICU admission were infections, especially respiratory infections and surgical site infections. A growing body of evidence supports that ICU stays are expensive, always occupy major hospital resources, and are associated with the worst outcomes. To date, there is insufficient evidence to determine which patients with digestive system tumors benefit the most from being admitted to the ICU after surgery. Therefore, this study intends to adopt retrospective study to determine the risk factors of postoperative ICU transfer for patients with digestive system malignant tumor, and build a risk prediction model for postoperative ICU admission, so as to guide the decision of postoperative ICU transfer for patients with digestive system malignant tumor.

DETAILED DESCRIPTION:
The incidence of malignant tumors of digestive system is increasing year by year in the world, and surgical treatment is the first choice for malignant tumors of digestive system. Most of these patients were elderly, had more complications before surgery, had greater surgical trauma, and had a high proportion of postoperative ICU admission. In recent three years, 28.1% of patients with malignant tumor of digestive system were admitted to ICU after surgery. The study found that postoperative ICU care in critically ill patients was conducive to reducing mortality, while non-essential postoperative ICU care in some patients was associated with the worst outcome. At present, there is still a lack of accurate and reliable decision making system for postoperative admission to ICU for patients with digestive system malignancies at home and abroad. Therefore, this project intends to establish a predictive model for postoperative ICU admission of patients with malignant tumors of the digestive system, develop a friendly interface that is convenient for medical care, help medical care quickly determine the biggest beneficiaries of postoperative ICU admission, rationally allocate medical resources, improve medical quality, reduce medical costs, ensure perioperative safety of patients, and promote postoperative rehabilitation of patients. At present, there is still a lack of accurate and reliable decision making system for postoperative admission to ICU for patients with digestive system malignancies at home and abroad. Therefore, this project intends to establish a predictive model for postoperative ICU admission of patients with malignant tumors of the digestive system, develop a friendly interface that is convenient for medical care, help medical care quickly determine the biggest beneficiaries of postoperative ICU admission, rationally allocate medical resources, improve medical quality, reduce medical costs, ensure perioperative safety of patients, and promote postoperative rehabilitation of patients.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients with malignant tumor of digestive system under general anesthesia, ASA Ⅱ~ Ⅳ

Exclusion Criteria:

* Emergency operation, operation stopped after entering the operating room, ASA > Ⅳ

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery for malignant tumors of digestive system under general anesthesia in Shaanxi Provincial Cancer Hospital and Ningxia Medical University General Hospital from January 2019 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
admitted to ICU after surgery | the day and three days after surgery
  whether the patient was admitted to ICU after surgery or within three days

CONTACTS AND LOCATIONS:
Overall Officials: Liqin Deng, M.D, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No